CLINICAL TRIAL: NCT03162822
Title: Targeting Parent-Child Coercion to Impact Health Behaviors and Regimen Adherence
Brief Title: Caregiver-Child Interaction and Health Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-01081; 1UH2DE025980-01 (NIH)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Early Childhood Caries; Caregiver-Child Coercion
Keywords: Caregiver-Child Coercion; Early Childhood Caries
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Within-subject design over 2 visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Intervention (Active Comparator): The cognitive intervention has parents come up with reasons why their children do things they don't like, until they come up with benign attributions for those behaviors.
  Interventions: Other: Cognitive Intervention
- Behavioral Intervention (Active Comparator): The behavioral intervention has the parents develop an if-then plan for dealing with conflict and negativity, using strategies to downregulate their own negative emotions.
  Interventions: Behavioral: Behavioral Intervention
- Interpretation Bias Intervention (Active Comparator): The Interpretation Bias intervention has parents look at "morphed" facial expressions and determine whether the face is happy or angry. Positive feedback is given for rating the faces as happy and negative feedback is given for rating the faces as angry.
  Interventions: Other: Interpretation Bias Intervention
- Evaluative Conditioning Intervention (Active Comparator): The Evaluative Conditioning intervention presents parents with pictures of ambiguous child faces (conditioned stimuli) and pairs them with positive word descriptors (unconditioned stimuli; e.g., sweet; cooperative).
  Interventions: Other: Evaluative Conditioning

INTERVENTIONS:
Behavioral: Behavioral Intervention — The behavioral intervention has the parents develop an if-then plan for dealing with conflict and negativity, using strategies to downregulate their own negative emotions.
  Arms: Behavioral Intervention
Other: Cognitive Intervention — The cognitive intervention has parents come up with reasons why their children do things they don't like, until they come up with benign attributions for those behaviors.
  Arms: Cognitive Intervention
Other: Interpretation Bias Intervention — The Interpretation Bias intervention has parents look at "morphed" facial expressions and determine whether the face is happy or angry. Positive feedback is given for rating the faces as happy and negative feedback is given for rating the faces as angry.
  Arms: Interpretation Bias Intervention
Other: Evaluative Conditioning — The Evaluative Conditioning intervention presents parents with pictures of ambiguous child faces (conditioned stimuli) and pairs them with positive word descriptors (unconditioned stimuli; e.g., sweet; cooperative).
  Arms: Evaluative Conditioning Intervention

SUMMARY:
Caregivers and their child are being asked to participate because the investigators are interested in typical caregiver-child interactions and health behaviors. In particular, the investigators are interested in different ways that caregivers react to and understand their young children's behavior, and their health behaviors.

DETAILED DESCRIPTION:
If they decide to participate in this study, caregivers and their child will come visit the laboratory twice at times that are convenient for them. The first visit will take 2.5-3 hours and the second visit will take 2-2.5 hours, so the subject runners will ask them to schedule them at times when their child will be well-rested and fed prior to arrival.

Here is a list of activities that the subject runners will ask caregivers and their child to participate in. These activities will be video-recorded and recordings will be kept digitally on a secure password-protected server. A separate consent form for the video-recording will be provided and caregivers must consent to the video-recording if they wish to participate in this study. Video-recordings will be assigned a random subject ID number.

* Upon arrival at the laboratory during both visits, the subject runners will explain the tasks to caregivers and the subject runners will set them and their child up with the machine that allows us to measure heart rate and skin moisture. This means the subject runners will place nine sensors on their and their child's bodies. These sensors will be placed on the collar bones, the lower left rib cage, the upper and mid-chest, the upper and midback, and the palm of their and their child's non-dominant hand. Caregivers and their child will still be able to move freely around the room.
* Next, the subject runners will either:

  * Conduct a short discussion where the subject runners will discuss caregivers' responses to their child's behavior or the intentions behind their child's behavior. A quarter of the research subjects in this study will complete a task where their responses to their child's behaviors are discussed and another quarter of the subjects will complete a task where the reasons for their child's behavior are discussed. Which type of discussion participants have will be "randomly assigned", which means that a computer will generate this decision before they arrive for their visit.
  * Or have caregivers complete a short computerized activity where caregivers will look at a series of images and descriptions or will be asked to rate a series of images with facial expressions. A quarter of the research subjects in this study will complete a computerized activity where they will look at a series of images and descriptions and another quarter of the subjects will complete a computerized activity where they will rate a series of images with facial expressions. Which type of activity participants have will be "randomly assigned", which means that a computer will generate this decision before they arrive for their visit.
* After this brief discussion, the subject runners will have caregivers and their child complete a series of tasks that are the sorts of activities they might encounter in daily life. In the first task the subject runners will have caregivers direct their child to clean up toys. In the second task the subject runners will have their child play with some toys while they are occupied on their phone. In the third task the subject runners will give them questionnaires to complete while their child waits on a mat. All three of these tasks will take 25-30 minutes.
* After this task, the subject runners will either:

  * Allow caregivers to have a break with their child. The subject runners will provide toys, drinks and snacks during the break. The subject runners will then ask caregivers to brush their child's teeth with a toothbrush that the subject runners provide, as they normally would.
  * Or have caregivers complete a task where they will rate what they felt and thought during their interaction with their child while watching a video of their interaction.
* At the end of these tasks the subject runners will provide caregivers with the opportunity to discuss the visit, their child's behaviors, and any other questions or concerns they may have. The subject runners will not ask them to participate in any additional visits or questionnaires after their second visit.

ELIGIBILITY:
Inclusion Criteria:

* Children between 18 and 36 months of age
* The primary caregiver of the child must be 18 years of age or older
* The primary caregiver must be the child's legal guardian
* The child in the dyad must have history of early childhood caries (ECC), have a sibling with a history of ECC, or be at risk for ECC
* The child in the dyad must qualify on behavioral problems

Exclusion Criteria:

-If individuals do not meet the above criteria, they will be excluded from the study.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Caregiver-Child Interaction Tasks | 30 Minutes per visit
  The subject runners will have caregivers and their child complete a series of tasks that are the sorts of activities they might encounter in daily life. In the first task the subject runners will have caregivers direct their child to clean up toys. In the second task the subject runners will have their child play with some toys while they are occupied on their phone. In the third task the subject runners will give them questionnaires to complete while their child waits on a mat.
Health Behaviors | 10 Minutes per visit
  Health Behaviors
Tooth brushing Task | 3 Minutes per visit
  The subject runners will ask caregivers to brush their child's teeth with a toothbrush that the subject runners provide, as they normally would.
Video-Mediated Emotion Recall | 30 Minutes per visit
  The video-mediated recall procedure (Gottman & Levenson, 1985; Lorber, 2007) is a procedure by which parents and/or a member of a couple view a videotape of their interaction with their partner or child. While watching the video, they use a dial to rate their experienced emotion and/or cognitions moment-by- moment during the interaction task.

SECONDARY OUTCOMES:
Psychophysiological Measures | 2-3 hours per visit
  The subject runners will set them and their child up with the machine that allows us to measure heart rate and skin moisture. This means the subject runners will place nine sensors on their and their child's bodies. These sensors will be placed on the collar bones, the lower left rib cage, the upper and mid-chest, the upper and midback, and the palm of their and their child's non-dominant hand. Caregivers and their child will still be able to move freely around the room.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Heyman, Ph.D., Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Smith Slep AM, Heyman RE, Mitnick DA, Lorber MF, Rhoades KA, Daly KA, Nichols SR, Eddy JM. Do Brief Lab-Based Interventions Decrease Coercive Conflict Within Couples and Parent-Child Dyads? Behav Ther. 2023 Jul;54(4):666-681. doi: 10.1016/j.beth.2023.01.006. Epub 2023 Feb 2. PMID 37330256

DOCUMENTS (1):
  • Informed Consent Form (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03162822/ICF_003.pdf